CLINICAL TRIAL: NCT06933810
Title: Examining the Ethical Attitudes of Nurses Working in a University Hospital
Status: Completed | Type: Observational
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Zeynal KİZİR, Principal Investigator, Hasan Kalyoncu University
Other Study IDs: HKU-SBF-KZ-01; HKU-SBF-KZ-01 (Other Grant/Funding Number: Hasan Kalyoncu University)
Record Dates: First submitted 2025-03-27; First posted 2025-04-18 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Ethics
Keywords: nursing; ethics; attitudes; nurse behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study aims to examine the ethical attitudes of nurses working in a university hospital.

The study includes nurses from departments such as internal medicine, surgery, intensive care, and emergency services.

A standardized data collection tool was used, and the study was conducted with volunteer participants.

This is a descriptive and cross-sectional observational study.

DETAILED DESCRIPTION:
This descriptive and cross-sectional study was conducted to evaluate the ethical attitudes of nurses working in a university hospital setting.

Nurses from various departments, including internal medicine, surgery, intensive care, and emergency services, participated in the study voluntarily.

Data were collected using the Nurse Information Form and the Ethical Attitudes in Nursing Care Scale.

The study aimed to gain insights into nurses' perceptions and behaviors related to ethical principles in clinical practice.

The findings are expected to contribute to the development of ethics training programs for nurses and to improve ethical standards in nursing care.

*No results or conclusions are included in this section, as required by ClinicalTrials.gov.*

ELIGIBILITY:
Inclusion Criteria:

* Nurses who are actively working in the hospital during the study period
* Nurses who agree to voluntarily participate in the study

Exclusion Criteria:

* Nurses who do not want to participate in the study
* Nurses who withdraw from the study at any stage

Ages: 21 Years to 51 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The population of the study consisted of a total of 690 nurses working in the internal medicine, surgery, intensive care, and emergency services of the hospital where the study was conducted. Without selecting a sample, nurses who were actively working between the specified dates and volunteered to participate in the study were included in the study. The entire population could not be reached because 50 nurses were on maternity leave and 133 nurses did not want to participate in the study. The study was completed with a total of 507 volunteer nurses, 144 of whom worked in internal medicine, 122 in surgery, 141 in intensive care, and 100 in emergency services.
Sampling Method: Non-Probability Sample
Enrollment: 507 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Nurses' Ethical Attitude Scores | Within 1 month from the date of data collection
  Total scores are calculated using the Ethical Attitudes in Nursing Care Scale. Score range: 15 (minimum) to 75 (maximum). Higher scores indicate more positive ethical attitudes among nurses.

CONTACTS AND LOCATIONS:
Overall Officials: NURAN TOSUN, PROF. DR., Study Director — HASAN KALYONCU UNIVERSİTY
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because I am the Responsible Author and will be following up the work myself.